CLINICAL TRIAL: NCT03185481
Title: A PHASE 2, OPEN LABEL EXTENSION STUDY TO INVESTIGATE THE LONG TERM SAFETY AND TOLERABILITY OF PF-06649751 IN SUBJECTS WITH MOTOR FLUCTUATIONS DUE TO PARKINSON'S DISEASE
Brief Title: Safety and Tolerability of PF-06649751 in Parkinson's Disease Patients With Motor Fluctuations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated 25Sep17 due to parent study insufficient efficacy. Not due to safety
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B7601017; 2017-000128-81 (EudraCT Number)
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Parkinson's Disease With Motor Fluctuations
Keywords: Parkinson's Disease; Motor Fluctuations; D1 partial agonist
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Depending on the actual treatment the subject received in B7601003, subjects will be randomized to one of 4 treatment groups (15 mg QD, 7 mg QD, 3 mg QD, or 1 mg QD group) and titrated up to 15 mg QD over a 3 week period, as appropriate.
  All subjects who were blindly down-titrated during the parent study (B7601003) will remain at/or be titrated to 7 mg QD only and remain at that dose for the rest of the B7601017 study in order to protect the blind for the parent study. Subjects who successfully titrate to 15 mg QD will enter the Adjustment Period at that dose. Subjects who cannot tolerate 15 mg QD at any time during the study will be allowed to down-titrate to 7 mg QD (but not lower) and will stay at that dose for the rest of the study. Subjects who cannot remain at a stable dose (7 mg or 15 mg QD) will be discontinued.
Who Masked: Participant, Care Provider, Investigator
Masking Description: During the titration phase, the allocation to treatment will be double blind to protect the blind of the parent study (B7601003). After completing the titration phase, the treatment assignment becomes open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- 1 mg QD to 15 mg QD PF-06649751 (Experimental): Up titration from 1 mg QD to 15 mg QD PF-06649751
  Interventions: Drug: 1 mg QD to 15 mg QD PF-06649751
- 3 mg QD to 15 mg QD PF-06649751 (Experimental): Up titration from 3 mg QD to 15 mg QD PF-06649751
  Interventions: Drug: 3 mg QD to 15 mg QD PF-06649751
- 7 mg QD to 15 mg QD PF-06649751 (Experimental): Up titration from 7 mg QD to 15 mg QD PF-06649751
  Interventions: Drug: 7 mg QD to 15 mg QD PF-06649751
- 15 mg QD PF-06649751 (Experimental): 15 mg QD PF-06649751 remains at 15 mg QD PF-06649751
  Interventions: Drug: 15 mg QD PF-06649751
- 1 mg to 7 mg QD PF-06649751 (Experimental): Up titration from 1 to 7 mg QD PF-06649751 if de-escalated in parent study
  Interventions: Drug: 1 mg QD to 7 mg QD PF-06649751 (if de-escalated in parent study)
- 3 mg QD to 7 mg QD PF-06649751 (Experimental): Up titration from 3 to 7 mg QD PF-06649751 if de-escalated in parent study
  Interventions: Drug: 3 mg QD to 7 mg QD PF-06649751 (de-escalated in parent study)
- 7 mg QD to 7 mg QD PF-06649751 (Experimental): 7 mg QD remains at 7 mg QD PF-06649751 if de-escalated in parent study
  Interventions: Drug: 7 mg QD to 7 mg QD PF-06649751 (de-escalated in parent study)
- 15 mg to 7 mg QD PF-06649751 (Experimental): 15 mg QD de-escalated to 7 mg QD in parent study B7601003 remain at 15 mg QD PF-06649751
  Interventions: Drug: 15 mg QD de-escalated to 7 mg QD PF-06649751 in parent study remain at 7 mg QD

INTERVENTIONS:
Drug: 1 mg QD to 15 mg QD PF-06649751 — Up titration from 1 mg QD to 15 mg QD PF-06649751
  Arms: 1 mg QD to 15 mg QD PF-06649751
Drug: 3 mg QD to 15 mg QD PF-06649751 — Up titration from 3 mg QD to 15 mg QD PF-06649751
  Arms: 3 mg QD to 15 mg QD PF-06649751
Drug: 7 mg QD to 15 mg QD PF-06649751 — Up titration from 7 mg QD to 15 mg QD PF-06649751
  Arms: 7 mg QD to 15 mg QD PF-06649751
Drug: 15 mg QD PF-06649751 — 15 mg QD PF-06649751 remaining at 15 mg QD PF-06649751
  Arms: 15 mg QD PF-06649751
Drug: 1 mg QD to 7 mg QD PF-06649751 (if de-escalated in parent study) — Up titration from 1 mg QD to 7 mg QD PF-06649751 for subject at 1 mg QD who were blindly de-escalated in the parent study
  Arms: 1 mg to 7 mg QD PF-06649751
Drug: 3 mg QD to 7 mg QD PF-06649751 (de-escalated in parent study) — Up titration from 3 mg QD to 7 mg QD PF-06649751 for 3 mg QD subjects who were blindly de-escalated in parent study
  Arms: 3 mg QD to 7 mg QD PF-06649751
Drug: 7 mg QD to 7 mg QD PF-06649751 (de-escalated in parent study) — 7 mg QD to remain at 7 mg QD PF-06649751 for subjects who were blindly de-escalated in parent study
  Arms: 7 mg QD to 7 mg QD PF-06649751
Drug: 15 mg QD de-escalated to 7 mg QD PF-06649751 in parent study remain at 7 mg QD — 7mg QD PF-06649751 for subjects assigned to 15 mg QD who were blindly de-escalated to 7 mg QD PF-06649751 in parent study
  Arms: 15 mg to 7 mg QD PF-06649751

SUMMARY:
The purpose of this study is to evaluate the long term safety and tolerability of PF-06649751 in Parkinson's disease patients who experience motor-fluctuations.

DETAILED DESCRIPTION:
This is an open label study evaluating the long term safety and tolerability of PF-06649751 in Parkinson's disease patients who experience motor-fluctuations. Subjects who completed Ph2 study B7601003 will be randomized to one of 4 treatment groups (15 mg QD, 7 mg QD, 3 mg QD, or 1 mg QD group) depending on the treatment received in B7601003 and titrated up to 15 mg QD over a 3 week period, as appropriate. All subjects who were blindly down-titrated during the B7601003 study will remain at/or be titrated to 7 mg QD only and remain at that dose for the rest of the B7601017 study in order to protect the blind for the prior study. Subjects who successfully titrate to 15 mg QD will enter the Adjustment Period at that dose.

Subjects who cannot tolerate 15 mg QD at any time during the study will be allowed to down-titrate to 7 mg QD (but not lower) and will stay at that dose for the rest of the study.

Subjects who cannot remain at a stable dose (7 mg or 15 mg QD) will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Having successfully completed parent study B7601003.
* Clinical diagnosis of Parkinson's disease.
* Able to refrain from any Parkinson's disease medication not permitted by the protocol.

Exclusion Criteria:

* Female of childbearing potential.
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality.
* Participation in other studies involving investigational drug(s), or treatment with any investigational drug within 30 days.

Ages: 40 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (9):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Associated Neurologists of Southern CT, PC, Fairfield, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Pharmaceutical Research Associates, Inc., Marlton, New Jersey
  - University of Toledo, Gardner-McMaster Parkinson Center, Toledo, Ohio
  - University of Toledo, Investigational Drug Services, Toledo, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Booth Gardner Parkinson's Care Center, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7601017&StudyName=Phase+2+Open+Label+Extension+Study+To+Investigate+The+Long+Term+Safety+And+Tolerability+Of+Pf-06649751
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7601017&StudyName=A+Phase+2+Open+Label+Extension+Study+To+Investigate+The+Long+Term+Safety+And+Tolerability+Of+Pf-06649751
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7601017&StudyName=A+Phase+2%2C+Open+Label+Extension+Study+To+Investigate+The+Long+Term+Safety+And+Tolerability+Of+Pf-06649751+In+Subjects+With+Motor+Fluctuations+Due+To+Parkinson%27s+Disease

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-06649751 15 mg: Participants who completed Week 15 in Study B7601003 (NCT02687542) were orally administered PF-06649751 once daily (QD) at the last dose level used in Study B7601003 (1 mg, 3 mg, 7 mg or 15 mg, and original placebo participants starting from 1 mg) titrated up to 15 mg during a 3-week titration period, followed by a 2-week dose adjustment period (15 mg or if intolerance, reduced to 7 mg) and then followed by open-label maintenance treatment of PF-06649751 15 mg QD for 44 weeks or until discontinuation.
Period: Overall Study
Arm/Group | PF-06649751 15 mg
Started | 5
Completed | 0
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Study Terminated by Sponsor | 4

BASELINE CHARACTERISTICS:
Arm/Group | PF-06649751 15 mg
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5
  Black or African American | 0
  Asian | 0
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  Other | 0
  Unknown | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (All Causalities)
Description: An adverse event (AE) is any untoward medical occurrence in a study participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. Any AE occurring following the start of treatment or occurring before treatment but increasing in severity afterward were counted as treatment-emergent AE (TEAE).
Time Frame: Baseline to last visit after termination (up to approximately 3 months)
Population: The study population included all participants who received at least 1 dose of study medication during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06649751 15 mg
Number analyzed (Participants) | 5
Participants | 3

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Treatment Related)
Description: An adverse event (AE) is any untoward medical occurrence in a study participant administered a product or medical device. Any AE occurring following the start of treatment or occurring before treatment but increasing in severity afterward were counted as treatment-emergent AE (TEAE).
Time Frame: Baseline to last visit after termination (up to approximately 3 months)
Population: The study population included all participants who received at least 1 dose of study medication during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06649751 15 mg
Number analyzed (Participants) | 5
Participants | 2

3. Primary Outcome: Number of Participants With Clinically Significant Findings in Physical Examination
Description: A full physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal and musculoskeletal systems. The clinical significance was determined by the investigator.
Time Frame: Baseline to last visit after termination (up to approximately 3 months)
Population: The study population included all participants who received at least 1 dose of study medication during the study period and had a post-baseline physical examination.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06649751 15 mg
Number analyzed (Participants) | 3
Participants | 0

4. Primary Outcome: Number of Participants With Clinically Significant Findings in Neurological Examination
Description: The full neurological examination included assessment of the visual fields and of the right and left optic fundus; cranial nerves; mental state; muscle strength and tone, abnormal movements; deep tendon reflexes; sensory exam, coordination, gait and station. Higher cortical and motor function was considered part of the complete neurological exam. The brief neurological exam included observation for cerebellar (intention) tremor and for non cerebellar tremors (eg, resting or positional), finger to nose, heel to shin, Romberg, gait and tandem walking, positional and gaze evoked nystagmus. The clinical significance was determined by the investigator.
Time Frame: Baseline to last visit after termination (up to approximately 3 months)
Population: The study population included all participants who received at least 1 dose of study medication during the study period and had a post-baseline neurological examination.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06649751 15 mg
Number analyzed (Participants) | 4
Participants | 0

5. Primary Outcome: Number of Participants With Abnormalities in Laboratory Test (Without Regard to Baseline Abnormality)
Description: Laboratory tests included hematology(hemoglobin,hematocrit,red and white blood cell count,mean corpuscular volume,mean corpuscular hemoglobin,mean corpuscular hemoglobin concentration,platelet count,neutrophils,eosinophils,monocytes, basophils,lymphocytes), chemistry(blood urea nitrogen/urea and creatinine,fasting glucose, calcium,sodium,potassium, chloride,total carbon dioxide,aspartate and alanine aminotransferase,total bilirubin,alkaline phosphatase,uric acid,albumin,total protein),urinalysis(pH,qualitative glucose protein,blood,ketones,nitrites,leukocyte esterase,urobilinogen,urine bilirubin,microscopy,specific gravity,urine creatinine),other tests(urine drug screen,follicle stimulating hormone,anti neutrophil cytoplasmic antibody panel,qualitative antinuclear antibody,fibrinogen,C reactive protein,erythrocyte sedimentation rate,C3, C4, CH50/CH100,rheumatoid factor,immunoglobulin panel,if anti- neutrophil cytoplasmic antibody positive:proteinase 3 Ab,myeloperoxidase Ab tests).
Time Frame: Baseline to last visit after termination(up to approximately 3 months)
Population: The study population included all participants who received at least 1 dose of study medication during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06649751 15 mg
Number analyzed (Participants) | 5
Participants | 1

6. Primary Outcome: Number of Participants With Vital Signs Data Meeting Pre-defined Criteria
Description: Number of participants with vital signs findings meeting the following criteria is presented:(1) standing DBP increase from baseline>= 20 mm Hg; (2) standing SBP increase from baseline>= 30 mm Hg; (3) supine DBP increase from baseline >=20 mm Hg; (4) supine SBP increase from baseline >=30 mm Hg; (5)standing DBP decrease from baseline>= 20 mm Hg; (6) standing SBP decrease from baseline>= 30 mm Hg; (7) supine DBP decrease from baseline >=20 mm Hg; (8) supine SBP decrease from baseline >=30 mm Hg.
Time Frame: Baseline to last visit after termination (up to approximately 3 months)
Population: The study population included all participants who received at least 1 dose of study medication during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06649751 15 mg
Number analyzed (Participants) | 5
Participants
  Standing DBP increase from baseline >= 20 mm Hg | 0
  Standing SBP increase from baseline >= 30 mm Hg | 1
  Supine DBP increase from baseline >= 20 mm Hg | 0
  Supine SBP increase from baseline >= 30 mm Hg | 2
  Standing DBP decrease from baseline >= 20 mm Hg | 0
  Standing SBP decrease from baseline >= 30 mm Hg | 0
  Supine DBP decrease from baseline >= 20 mm Hg | 0
  Supine SBP decrease from baseline >= 30 mm Hg | 0

7. Primary Outcome: Number of Participants With Vital Signs Data of Orthostatic Hypotension Meeting Pre-defined Criteria
Description: Orthostatic hypotension was defined as a decrease of >=20 mmHg for systolic blood pressure (SBP) or >=10 mmHg for diastolic blood pressure (DBP) 2 minutes after standing from a supine position.
Time Frame: Baseline to last visit after termination (up to approximately 3 months)
Population: The study population included all participants who received at least 1 dose of study medication during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06649751 15 mg
Number analyzed (Participants) | 5
Participants
  DBP postural difference>=10 mm Hg(Supine-Standing) | 3
  SBP postural difference>=20 mm Hg(Supine-Standing) | 4

8. Primary Outcome: Number of Participants With Electrocardiogram Data Meeting Pre-defined Criteria
Description: PR interval (time from the beginning of P wave to the start of QRS complex, corresponding to the end of atrial depolarization and onset of ventricular depolarization), QRS duration (time from Q wave to the end of S wave, corresponding to ventricle depolarization), QT interval (time from the beginning of Q wave to the end of T wave) and QTcF interval ( QT interval corresponding to electrical systole corrected for heart rate using Fridericia's formula) are summarized. Number of participants with ECG findings meeting the following criteria is presented: (1) PR interval >=300 msec; (2) QRS duration >=140 msec; (3) QT interval >= 500; (4) QTcF interval: 450 to <480 msec; (5) QTcF interval: 480 to <500 msec; (6) QTcF interval >=500 msec.
Time Frame: Baseline to last visit after termination (up to approximately 3 months)
Population: The study population included all participants who received at least 1 dose of study medication during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06649751 15 mg
Number analyzed (Participants) | 5
Participants
  PR Interval (aggregate) >= 300 msec | 0
  QRS Duration (aggregate) >= 140 msec | 0
  QT Interval (aggregate) >= 500 msec | 0
  QTcF Interval (aggregate) >= 450 msec, <480msec | 0
  QTcF Interval (aggregate) >= 480 msec, <500msec | 0
  QTcF Interval (aggregate) >= 500 msec | 0

9. Primary Outcome: Number of Participants With Worsening Suicidality and New Onset Suicidality
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) is an interview based rating scale to systematically assess suicidal ideation and suicidal behavior. At each suicidality assessment, participants felt to have significant suicidal ideation with actual plan and intent or suicidal behavior, must be evaluated by a clinician/mental health professional (MHP) skilled in the evaluation of suicidality in the participants by virtue of training or experience who determined if it is safe for the participants to participate/continue in the trial. The denominator used in the percentages was the number of participants assessed for suicidality or worsening, the denominator included the subset of participants who had any level of suicidality reported at baseline. For new onset, the denominator included the subset of participants with no suicidality reported at baseline.
Time Frame: Baseline to last visit after termination (up to approximately 3 months)
Population: The study population included all participants who received at least 1 dose of study medication during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06649751 15 mg
Number analyzed (Participants) | 5
Participants
  New Onset | 0
  Worsening | 0

10. Primary Outcome: Number of Participants With Benzodiazepine Discontinuation Symptoms Based on Physician Withdrawal Checklist (PWC-20)
Description: The PWC-20 is a physician-completed, 20-item reliable and sensitive instrument for the assessment of benzodiazepine discontinuation symptoms, including anxiety and nervous, depersonalization and derealization, diarrhea, diaphoresis, difficulty concentrating and remembering, dizziness-lightheadedness, depression, fatigue, lethargy and lack of energy, headaches, increased acuity for sound, smell, touch, or pain, insomnia, irritability, loss of appetite, muscle aches or stiffness, nausea-vomiting paresthesias, poor coordination, restlessness and agitation, tremor-tremulousness, and weakness. Summaries of the count of participants experiencing symptoms and severity listed in the PWC-20 were provided.
Time Frame: At last visit
Population: The population for PWC-20 included participants who completed study treatment and who participated the first visit of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06649751 15 mg
Number analyzed (Participants) | 4
Participants
  Anxiety, Nervousness: Not Present | 3
  Anxiety, Nervousness: Mild | 1
  Anxiety, Nervousness: Moderate | 0
  Anxiety, Nervousness: Severe | 0
  Difficult Concentrating, Remembering: Not Present | 3
  Difficult Concentrating, Remembering: Mild | 1
  Difficult Concentrating, Remembering: Moderate | 0
  Difficult Concentrating, Remembering: Severe | 0
  Dysphoric Mood, Depression: Not Present | 3
  Dysphoric Mood, Depression: Mild | 1
  Dysphoric Mood, Depression: Moderate | 0
  Dysphoric Mood, Depression: Severe | 0
  Fatigue, Lethargy, Lack of Energy: Not Present | 2
  Fatigue, Lethargy, Lack of Energy: Mild | 1
  Fatigue, Lethargy, Lack of Energy: Moderate | 1
  Fatigue, Lethargy, Lack of Energy: Severe | 0
  Insomnia: Not Present | 2
  Insomnia: Mild | 1
  Insomnia: Moderate | 1
  Insomnia: Severe | 0
  Irritability: Not Present | 3
  Irritability: Mild | 0
  Irritability: Moderate | 1
  Irritability: Severe | 0
  Muscle Aches or Stiffness: Not Present | 3
  Muscle Aches or Stiffness: Mild | 0
  Muscle Aches or Stiffness: Moderate | 1
  Muscle Aches or Stiffness: Severe | 0
  Poor Coordination: Not Present | 2
  Poor Coordination: Mild | 1
  Poor Coordination: Moderate | 1
  Poor Coordination: Severe | 0
  Restlessness, Agitation: Not Present | 3
  Restlessness, Agitation: Mild | 0
  Restlessness, Agitation: Moderate | 1
  Restlessness, Agitation: Severe | 0
  Tremor-Tremulousness: Not Present | 3
  Tremor-Tremulousness: Mild | 0
  Tremor-Tremulousness: Moderate | 0
  Tremor-Tremulousness: Severe | 1
  Weakness: Not Present | 2
  Weakness: Mild | 2
  Weakness: Moderate | 0
  Weakness: Severe | 0

11. Secondary Outcome: Change From Baseline for Hauser Participant Diary Data in Daily OFF Time
Description: Available diaries are designed to record participant motor state for half hour intervals. These diaries are a way for participant to assess their own health status without clinician bias or interpretation. In participant diaries, "OFF" time is defined as a period when medication has worn off and is no longer providing benefit with regard to mobility, slowness, and stiffness. During this period, Parkinson's Disease (PD) participants experience relatively poor overall function with worsening of tremor, rigidity, balance, or bradykinesia.
Time Frame: Baseline, Day 21 and Day 35
Population: The study population included all participants who received at least 1 dose of study medication during the study period.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | PF-06649751 15 mg
Number analyzed (Participants) | 1
Hours
  Baseline | 3.25 (NA) — As only 1 participant was analyzed, the calculation for standard deviation was not available.
  Day 21 | 0.00 (NA) — As only 1 participant was analyzed, the calculation for standard deviation was not available.
  Day 35 | -0.42 (NA) — As only 1 participant was analyzed, the calculation for standard deviation was not available.

12. Secondary Outcome: Change From Baseline for Hauser Participant Diary Data in Daily ON Time With Troublesome Dyskinesia
Description: Available diaries are designed to record participant motor state for half hour intervals. These diaries are a way for participants to assess their own health status without clinician bias or interpretation. "ON" time is defined as the time when medication is providing benefit with regard to mobility, slowness, and stiffness. "ON" time can be classified as associated with or without troublesome dyskinesia that interfere with activities of daily living.It has been demonstrated that "ON" time with troublesome dyskinesia are generally considered by participants to be "bad time" with regard to motor function.
Time Frame: Baseline, Day 21 and Day 35
Population: The study population included all participants who received at least 1 dose of study medication during the study period.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | PF-06649751 15 mg
Number analyzed (Participants) | 1
Hours
  Baseline | 0.00 (NA) — As only 1 participant was analyzed, the calculation for standard deviation was not available.
  Day 21 | 0.00 (NA) — As only 1 participant was analyzed, the calculation for standard deviation was not available.
  Day 35 | 0.00 (NA) — As only 1 participant was analyzed, the calculation for standard deviation was not available.

13. Secondary Outcome: Change From Baseline for Hauser Participant Diary Data in Daily ON Time Without Troublesome Dyskinesia
Description: Available diaries are designed to record participant motor state for half hour intervals. These diaries are a way for participants to assess their own health status without clinician bias or interpretation. "ON" time is defined as the time when medication is providing benefit with regard to mobility, slowness, and stiffness. "ON" time can be classified as associated with or without troublesome dyskinesia that interfere with activities of daily living. "ON" time without dyskinesia and on time with non troublesome dyskinesia are generally considered to be "good time".
Time Frame: Baseline, Day 21 and Day 35
Population: The study population included all participants who received at least 1 dose of study medication during the study period.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | PF-06649751 15 mg
Number analyzed (Participants) | 1
Hours
  Baseline | 9.58 (NA) — As only 1 participant was analyzed, the calculation for standard deviation was not available.
  Day 21 | 1.17 (NA) — As only 1 participant was analyzed, the calculation for standard deviation was not available.
  Day 35 | 2.42 (NA) — As only 1 participant was analyzed, the calculation for standard deviation was not available.

14. Secondary Outcome: Change From Baseline in Movement Disorder Society Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I, II, III, IV, and Total Score
Description: The total MDS-UPDRS score developed by the Movement Disorder Society is the most common method of evaluating the severity of Parkinson's Disease (PD). Part I assesses non motor experiences of daily living(range 0-52).Part II assesses motor experiences of daily living(0-52). Part III assesses the motor signs of PD.Part IV assesses motor complications, dyskinesias, and motor fluctuations(0-24).Total Score:The sum of Parts I, II, III, and IV.Each question is anchored with five responses:0=normal, 1=slight, 2=mild, 3= moderate, 4=severe.Higher part and total scores indicate more severe signs of PD.There are four subscales in Part III:the tremor subscale(range 0-36),the rigidity subscale(0-20),the bradykinesia subscale(0-36),the postural instability and gait disorder (PIGD) subscale(0-12).
Time Frame: Baseline to last visit after termination (up to approximately 3 months)
Population: The study population included all participants who received at least 1 dose of study medication during the study period.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | PF-06649751 15 mg
Number analyzed (Participants) | 5
Units on a scale
  Part I Score | -1.5 [-15 to 9]
  Part II Score | 0 [-10 to 9]
  Part III Score | -2.5 [-9 to 11]
  Part IV Score | 0 [-3 to 6]
  Total Score | 0 [-32 to 19]

ADVERSE EVENTS:
Time Frame: Baseline to last visit after termination (up to approximately 3 months)
Arm/Group | PF-06649751 15 mg
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06649751 15 mg (N=5)
Hip Fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06649751 15 mg (N=5)
Fall (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 2
Orthostatic hypotention (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
This study was early terminated,not due to safety concern,but lack of sufficient demonstrated efficacy of the study drug to improve PD symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/81/NCT03185481/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT03185481/SAP_001.pdf